CLINICAL TRIAL: NCT00611806
Title: A Placebo-Controlled Trial of Folate With B12 in Schizophrenia Patients With Residual Symptoms
Brief Title: Effectiveness of Vitamin Supplementation in Treating People With Residual Symptoms of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH070831 (NIH); R01MH070831 (NIH); DATR A5-ETPD
Record Dates: First submitted 2008-02-07; First posted 2008-02-11 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: Cognition; Folic Acid; B12
MeSH Terms: conditions — Schizophrenia | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folate with B12 (Active Comparator): Participants will take folic acid plus B12 for 18 weeks.
  Interventions: Dietary Supplement: Folic Acid; Dietary Supplement: B12
- Placebo (Placebo Comparator): Participants will take placebo for 18 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Folic Acid — Folic acid 2mg po daily
  Arms: Folate with B12
Dietary Supplement: B12 — B12 400 micrograms po daily
  Other Names: cobalamin
  Arms: Folate with B12
Other: Placebo — 1 capsule po daily
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of folate and B12 supplementation in reducing negative symptoms in people with schizophrenia.

DETAILED DESCRIPTION:
About 30% of people with schizophrenia suffer from treatment-resistant psychotic symptoms, which may include social withdrawal, apathy, and depression. These negative symptoms can produce substantial distress for those affected, often disrupting social and occupational functioning and resulting in hospitalization. Although atypical antipsychotic medications have demonstrated some success in treating negative symptoms, the degree to which many negative symptoms respond is unclear. Depression and poor response to antidepressant medication have been linked to deficiency in the vitamins folate and B12. It is believed that vitamin supplementation with folate and B12 may offer a safe and inexpensive approach to improve outcomes for people with schizophrenia who have residual negative symptoms and have exhibited poor treatment response. This study will compare the effectiveness of folate and B12 versus placebo in reducing negative symptoms in people with schizophrenia.

Participation in this double-blind study will last 19 weeks. Potential participants will undergo initial screening, which will include a medical and psychiatric evaluation, physical exam, blood draw, urine sampling, and questionnaires. Participants will also be asked for permission to use a portion of the blood sample for genetic analysis. Eligible participants will be randomly assigned to take folate with B12 or placebo. Participants will first complete a 2-week stabilization phase, followed by the 16-week treatment study. Medication visits, occurring every 2 weeks during treatment, will include questions about medication side effects and the distribution of study medication. During specified medication visits, participants will complete various assessments, which will include questionnaires about schizophrenia, tests of learning and memory, repeat blood tests, and pregnancy tests. The medication visits will last between 15 minutes and 4 hours, depending on the scheduled assessments for that visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, any subtype
* Treated with an antipsychotic medication for at least 6 months at a stable dose for at least 6 weeks before study entry
* PANSS total score of at least 60, with a score of at least 3 (moderate) on one negative symptom item or on one positive symptom item
* Simpson Angus Scale (SAS) for Extrapyramidal Syndrome (EPS) total score of 12 or less
* A score of 2 (mild) or less on all items of the Calgary Depression Scale (CDS)
* Speaks English adequately enough to complete cognitive testing

Exclusion Criteria:

* Serum B12 concentration less than 300 ug/L
* Complete blood count results consistent with megaloblastic anemia
* Serum creatinine concentration greater than 1.4
* Current use of folate or B12 supplementation
* Current use of any of the following medications: phenobarbital, phenytoin, carbamazepine, valproic acid, fosphenytoin, primidone, or pyrimethamine
* Alcohol or other substance abuse within 3 months before study entry (nicotine allowed)
* Positive baseline urine toxic screen
* Unstable medical illness
* Unstable psychiatric illness
* Seizure disorder
* Pregnant or breastfeeding

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital Schizophrenia Program - Freedom Trail Clinic, Boston, Massachusetts
  - Touchstone innovare, Grand Rapids, Michigan
  - URMC Severe Mental Disorders Program, Rochester, New York

REFERENCES:
- [Result] Roffman JL, Lamberti JS, Achtyes E, Macklin EA, Galendez GC, Raeke LH, Silverstein NJ, Smoller JW, Hill M, Goff DC. Randomized multicenter investigation of folate plus vitamin B12 supplementation in schizophrenia. JAMA Psychiatry. 2013 May;70(5):481-9. doi: 10.1001/jamapsychiatry.2013.900. PMID 23467813

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 189 Participants were screened for enrollment, but 49 were excluded. 40 were ineligible, 2 withdrew consent, 1 terminated because of an adverse event, and 6 were terminated because of study visit noncompliance.
Period: Overall Study
Arm/Group | Folate With B12 | Placebo
Started | 94 | 46
Completed | 78 | 43
Not Completed | 16 | 3
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Folate With B12 | Placebo | Total
Number analyzed (Participants) | 94 | 46 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.3 (1.1) | 45.9 (1.6) | 45.6 (1.35)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 46 | 140
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 66 | 14 | 80
Region of Enrollment [Number; unit: participants]
  United States | 94 | 46 | 140

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The change from baseline on the Positive and Negative Syndrome Scale (PANSS).The PANNS has three subscales: positive (score range 7-49), negative (score range 7-49), and general psychopathology (score range 16-112). The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7, representing positive symptoms of schizophrenia. The PANSS negative symptom subscale is comprised of 7 items rated on a scale of 1-7 representing the negative symptoms of schizophrenia, and the general psychopathology subscale is comprised of 16 items rated on a scale of 1-7 representing symptoms of general psychopathology in mental illness. The total score was computed by adding all the items on the sub-scale together. Scores reported are change in symptoms per week, relative to baseline. A negative score represents a decrease in total PANSS score per week, whereas a positive score represents an increase in total PANSS score per week.
Time Frame: Baseline vs. Week 16
Population: Participants analyzed were those who completed at least 1 post-baseline visit or more (n = 135). 120 participants completed the study to the week 16 endpoint; however, 15 participants did not complete the entire 16 weeks, but completed at least one post-baseline study visit where the PANSS assessment was performed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Folate With B12 | Placebo
Number analyzed (Participants) | 89 | 46
units on a scale | -.21 [-.35 to -.07] | -.22 [-.42 to -.03]

2. Secondary Outcome: Cognitive Deficits, as Measured by the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Cognitive Battery Composite Score
Time Frame: Measured at Week 16
Reporting Status: Not Posted

3. Secondary Outcome: Positive Sub Scale of the Positive and Negative Syndrome Scale (PANSS)
Description: The change from baseline on the positive symptom sub-scale of the Positive and Negative Syndrome Scale (PANSS). Total PANSS positive symptom sub-scale scores range from 7-49. The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. A score of one on each item 1 absent, 2 is minimal, 3 is mild, 4 is moderate, 5 is moderately severe, 6 is severe, and 7 is extreme. The total score was computed by adding all the items on the sub-scale together. Scores reported are change in symptoms per week, relative to baseline. A negative score represents a decrease in total PANSS score per week, whereas a positive score represents an increase in total PANSS score per week.
Time Frame: Baseline vs. Week 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Folate With B12 | Placebo
Number analyzed (Participants) | 89 | 46
units on a scale | -.06 [-.12 to -.01] | -.04 [-.11 to .03]

4. Secondary Outcome: Scale for Assessment of Negative Symptoms (SANS)
Description: The change from baseline on the scale for the assessment of negative symptoms (SANS) total score. Total SANS scores range from 0-100. The SANS is comprised of 5 subscores: Affective Flattening or Blunting (score range 0-35), Alogia (score range 0-20), Avolition-Apathy (score range 0-15), Anhedonia-Asociality (score range 0-20), and Attention (0-10). For each scale, the higher the score the more prominent the negative symptoms were. The total score was computed by adding all the sub-scale total scores. Scores reported are change in symptoms per week, relative to baseline. A negative score represents a decrease in total SANS score per week, whereas a positive score represents an increase in total SANS score per week.
Time Frame: Baseline vs. Week 16
Population: Participants analyzed were those who completed at least 1 post-baseline visit or more (n = 135). 120 participants completed the study to the week 16 endpoint; however, 15 participants did not complete the entire 16 weeks, but completed at least one post-baseline study visit where the SANS assessment was performed.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Folate With B12 | Placebo
Number analyzed (Participants) | 89 | 46
units on a scale | -.19 [-.35 to -.03] | .02 [-.21 to .24]

5. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) and FOLH1, MTHRF, MTR, and COMT Genotype
Description: The change from baseline on the Positive and Negative Syndrome Scale (PANSS) (including FOLH1, MTHRF, MTR, and COMT genotype simultaneously into a linear mixed model).The PANNS has three sub-scales: positive (score range 7-49), negative (score range 7-49), and general psychopathology (score range 16-112). The PANSS negative and positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7 representing the negative and positive symptoms of schizophrenia, respectively, and the general psychopathology sub-scale is comprised of 16 items rated on a scale of 1-7 representing symptoms of general psychopathology in mental illness. The total score was computed by adding all the items on the sub-scale together. Scores reported are change in symptoms per week, relative to baseline. A negative score represents a decrease in total PANSS score per week, whereas a positive score represents an increase in total PANSS score per week.
Time Frame: Baseline vs. Week 16
Population: Participants analyzed were those who completed at least 1 post-baseline visit or more (n = 135) and agreed to the DNA blood draw (n = 120).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Folate With B12 | Placebo
Number analyzed (Participants) | 79 | 41
units on a scale | -.21 [-.35 to -.07] | -.1 [-.31 to .11]

6. Secondary Outcome: Relationship Between Response of Negative and Positive Symptoms and the Change in RBC Folate, Serum Folate, Serum B12, and Plasma Homocysteine Concentrations
Time Frame: Measured at Week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Folate With B12 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/94 | 4/46
Other Adverse Events (participants affected / at risk) | 21/94 | 16/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folate With B12 (N=94) | Placebo (N=46)
Hospitalization due to worsening psychosis (Psychiatric disorders) | 1 (2) | 1 (2)
Cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Body Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal Tendency (Psychiatric disorders) | 1 (1) | 0 (0)
Vision Decreased (Eye disorders) | 0 (0) | 1 (1)
Brain Tumor (Nervous system disorders) | 0 (0) | 1 (1)
Irritation of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Folate With B12 (N=94) | Placebo (N=46)
Constipation (Nervous system disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Cholelithiasis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dirrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1) | 0 (0)
Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Delusions (Psychiatric disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Injury (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Manic Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Muscle Spasm (Nervous system disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Suicidal Tendency (Psychiatric disorders) | 1 (1) | 0 (0)
Back Pain (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Eye Blood Shot (Eye disorders) | 0 (0) | 1 (1)
Vision Decreased (Eye disorders) | 0 (0) | 1 (1)
Asthema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Brain Tumor (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Laboratory Test Abnormality (General disorders) | 1 (1) | 0 (0)
Irritation of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No